CLINICAL TRIAL: NCT00002427
Title: A Phase I/II Study of the Safety and Antiretroviral Activity of Nine Hydroxyurea Regimens in Combination With ddI and d4T in Subjects With HIV Infection
Brief Title: Safety and Effectiveness of Combining Hydroxyurea (HU) With Didanosine (ddI) and Stavudine (d4T) for Treatment of HIV-Infected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Research Institute for Genetic and Human Therapy (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Factorial | Purpose: Treatment
Other Study IDs: 304A; RIGHT 702
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-08

CONDITIONS: HIV Infections
Keywords: Didanosine; Dose-Response Relationship, Drug; Drug Therapy, Combination; Stavudine; Hydroxyurea; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Hydroxyurea; Stavudine; Didanosine

INTERVENTIONS:
Drug: Hydroxyurea
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of 9 doses of HU in order to find the best dose of HU to use with ddI and d4T in fighting HIV infection.

HU plus ddI plus d4T appears to be a suitable anti-HIV drug combination for long-term control of HIV. This combination can sharply decrease viral load (level of HIV in the body) with few side effects, making it easy to take.

DETAILED DESCRIPTION:
The combination of HU plus ddI plus d4T appears to be suitable for long-term control of HIV in that it: (1) has a novel resistance/rebound profile demonstrating virus suppression even in the presence of ddI-resistant mutants; (2) can produce a pronounced fall in viral load; and (3) is well tolerated (over 200 patients have been treated for up to 3 years with minimal side effects).

Patients are stratified by antiretroviral experience: naive (no more than 2 weeks of therapy) versus experienced (more than 2 weeks). Patients must discontinue all antiretroviral therapy for at least 28 days prior to randomization to 1 of 9 HU treatment arms. Treatment arms are divided into 3 HU dose categories: very low, low, and medium. Within each category HU is administered daily on 3 different dosing schedules. Depending on viral load, patients on the very low and low dose arms may have the opportunity to intensify their HU dose at any time beyond Week 12, provided no Grade 3 or 4 HU-related toxicity is present (these patients are monitored for an additional 8 weeks following intensification). All patients receive ddI and d4T at the same doses every day. When 50% of patients have completed 24 weeks of treatment, an analysis is made to determine whether or not to continue the 52-week study without modifications. Patients are monitored periodically for changes in plasma HIV RNA, CD4 cell counts, weight, and symptoms.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a viral load of 5,000 to 100,000 copies/ml.
* Are willing to stop all anti-HIV medications for at least 28 days before receiving study drugs.
* Are at least 18 years old.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a history of opportunistic (AIDS-related) infection.
* Have a history of pancreatitis or other serious condition.
* Have any cancer that will require chemotherapy within the next 24 weeks.
* Are allergic to ddI or d4T.
* Have received an HIV vaccine within 28 days of study entry.
* Have received a red blood cell transfusion within the past 60 days, or have had repeated transfusions at any time in the past.
* Abuse alcohol or drugs.
* Have received certain medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225
Dates: Start 1999-05

CONTACTS AND LOCATIONS:
Overall Officials: Franco Lori, Study Chair; Julianna Lisziewicz, Study Chair
Locations (18):
- United States (18):
  - AIDS Healthcare Foundation, Los Angeles, California
  - San Francisco VA Med Ctr, San Francisco, California
  - Gary Blick MD, Stamford, Connecticut
  - Dr Bruce Rashbaum, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Boulevard Comprehensive Care Ctr, Jacksonville, Florida
  - Center for Quality Care, Tampa, Florida
  - AIDS Research Consortium of Atlanta Inc, Atlanta, Georgia
  - New England Med Ctr, Boston, Massachusetts
  - Albany Med College, Albany, New York
  - Mt Vernon Hosp, Mount Vernon, New York
  - Univ of Pennsylvania Med Ctr, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ, Philadelphia, Pennsylvania
  - Coastal Carolina Research Ctr, Mt. Pleasant, South Carolina
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Texas Med Branch, Galveston, Texas
  - Montrose Clinic, Houston, Texas
  - Swedish Med Ctr, Seattle, Washington